CLINICAL TRIAL: NCT06832943
Title: A Prospective Multicenter Single-Arm Trial Evaluating the Efficacy and Safety of Robotic Bronchoscopy System-Assisted Stent Placement in Patients with Malignant Central Airway Stenosis
Brief Title: The Efficacy and Safety of Robotic Bronchoscopy System-Assisted Stent Placement in Patients with Malignant Central Airway Stenosis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Guangzhou Medical University (Other)
Responsible Party: Principal Investigator, Li Shiyue, Professor, Guangzhou Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RBS-Stent
Record Dates: First submitted 2025-02-12; First posted 2025-02-18 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-02

CONDITIONS: Airway Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- RBS group (Experimental): Patients with airway stenosis undergo stent placement with the help of RBS.
  Interventions: Procedure: Unicorn system

INTERVENTIONS:
Procedure: Unicorn system — Patients with airway stenosis undergo stent placement with the help of RBS.

SUMMARY:
The primary aim of this research is to assess the efficacy and safety of the bronchial navigation positioning equipment in assisting stent implantation for malignant central airway stenosis while guaranteeing the safety of the participants and the scientificity of the clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Patients are eligible only if they fulfill all of the following criteria:

  1. Age ≥ 18 years, regardless of gender;
  2. Patients voluntarily consent to airway stent implantation and meet the requirements for airway stent implantation under general anesthesia;
  3. Confirmed as having malignant central airway stenosis through bronchoscopy and being ineligible for surgery or refusing surgery, and in need of airway stent implantation.

Patients should be able to understand the purpose of the trial, demonstrate good compliance with the examinations and follow-ups, and voluntarily participate in the clinical trial and sign the informed consent form.

Exclusion Criteria:

* Patients fulfilling any of the following criteria will be excluded from this study:

  1. Severe dysfunction of the heart, lungs, liver, or kidneys, intolerant of bronchoscopic treatment;
  2. Apparent coagulation dysfunctions;
  3. Pregnant or lactating women, or participants with a pregnancy plan during the study period;
  4. Patients with implanted cardiac pacemakers, implanted defibrillators, or other active implants;
  5. Participants allergic to photosensitizers or anesthetics, or with a history of multiple severe allergies or hereditary allergies;
  6. Participants who have participated in or are currently participating in drug clinical trials within the past 3 months, or in other medical device clinical trials within the past 30 days; Other circumstances that the investigator considers inappropriate for participation in this clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-02-15 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
The success rate of stent placement | During the bronchoscopy
  The success rate of stent placement = (The number of patients with successful stent placement / The number of patients undergoing stent placement surgery) × 100% Successful placement: The stent is placed in the appropriate position without displacement, and the upper and lower ends of the stent are unobstructed.

IPD SHARING:
Plan to Share IPD: No